CLINICAL TRIAL: NCT00642330
Title: Randomized Pilot Study Comparing Oral Ibuprofen With Intravenous Ibuprofen in Very Low Birth Weight Infants With Patent Ductus Arteriosus
Brief Title: Comparative Study of Efficacy and Safety of Oral Ibuprofen and Intravenous Ibuprofen in Closure of Patent Ductus Arteriosus in Very Low Birth Weight Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital La Rabta (Other)
Collaborators: maternity and neonatal center (Unknown)
Responsible Party: khrouf naima, Hopital La Rabta
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IBU-001; TIS-1447; FMND-4585
Record Dates: First submitted 2008-03-17; First posted 2008-03-25 (Estimated); Last update posted 2008-03-25 (Estimated); Status verified 2008-03

CONDITIONS: Patent Ductus Arteriosus
Keywords: patent; ductus; arteriosus; ibuprofen; premature; infant
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator)
  Interventions: Drug: intravenous ibuprofen
- O (Active Comparator)
  Interventions: Drug: oral ibuprofen

INTERVENTIONS:
Drug: oral ibuprofen — one (10 mg / kg), two (10 mg / kg followed 24 hours after by 5 mg /kg) or three (10 mg / kg followed at 24-hour intervals by two doses of 5 mg /kg each) doses of oral ibuprofen starting on the third day of life.the number of doses is depending on echocardiographic findings concerning ductal closure.
  Arms: O
Drug: intravenous ibuprofen — one (10 mg / kg), two (10 mg / kg followed 24 hours after by 5 mg /kg) or three (10 mg / kg followed at 24-hour intervals by two doses of 5 mg /kg each) doses of oral ibuprofen starting on the third day of life.the number of doses is depending on echocardiographic findings concerning ductal closure.
  Arms: I

SUMMARY:
it is a prospective randomized simple-blinded pilot trial with the principal aim to compare efficacy and tolerance between oral ibuprofen and intravenous ibuprofen in early curative closure of PDA in very low birth weight infants. The likelihood of ductal closure with only one or two doses of treatment is a secondary objective.

DETAILED DESCRIPTION:
We calculated that a study group of 62 patients would be necessary for the study to be able to detect a difference of at least 25 percentage points in the closure rate between the oral ibuprofen and intravenous ibuprofen groups, assuming a closure rate of 65 percent with intravenous ibuprofen, with a p value of 0, 05 and a power of 80 percent.Patients (gestational age, 25 to 32 weeks) with echocardiographically confirmed patent ductus arteriosus and respiratory distress will randomly be assigned to receive one (10 mg / kg), two (10 mg / kg followed 24 hours after by 5 mg /kg) or three (10 mg / kg followed at 24-hour intervals by two doses of 5 mg /kg each) doses of either intravenous ibuprofen (group I, n = 32) or oral ibuprofen (group O, n = 32), starting on the third day of life. The rate of ductal closure, side effects, complications, and the patients' clinical course will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* a gestational age < 32 weeks
* a birth weight < 1500g
* a postnatal age between 48 and 96 hours, a respiratory distress requiring more than 25 % of oxygen supplementation
* an echocardiographic evidence of left to right significant shunting PDA

Exclusion Criteria:

* a right-to-left shunting
* major congenital anomalies
* IVH grade 3-4
* a tendency to bleed (defined by the presence of blood in the endotracheal aspirate, gastric aspirate, stools or urines and / or oozing from puncture sites)
* a serum creatinine level >140µmol/l, a serum urea nitrogen > 14 µmol/l and a platelet count < 60000/mm3.

Ages: 48 Hours to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
rate of ductal closure

SECONDARY OUTCOMES:
rate of side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Maternity and Neonatal Center, Tunis, Tunisia

REFERENCES:
- [Result] Cherif A, Jabnoun S, Khrouf N. Oral ibuprofen in early curative closure of patent ductus arteriosus in very premature infants. Am J Perinatol. 2007 Jun;24(6):339-45. doi: 10.1055/s-2007-981853. Epub 2007 Jun 12. PMID 17564958
- [Derived] Cherif A, Khrouf N, Jabnoun S, Mokrani C, Amara MB, Guellouze N, Kacem S. Randomized pilot study comparing oral ibuprofen with intravenous ibuprofen in very low birth weight infants with patent ductus arteriosus. Pediatrics. 2008 Dec;122(6):e1256-61. doi: 10.1542/peds.2008-1780. PMID 19047225